CLINICAL TRIAL: NCT02238262
Title: Observation of Therapy With Micardis® (Telmisartan) in Patients With Essential Hypertension in Hospitals
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.374
Record Dates: First submitted 2014-09-11; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- essential hypertension patients
  Interventions: Drug: Telmisartan

INTERVENTIONS:
Drug: Telmisartan
  Other Names: Micardis®; low and high dose

SUMMARY:
The aim of the observational study was to supplement the data on efficacy, safety and tolerability of telmisartan under daily conditions in hospitals

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of essential hypertension
* Minimum age of 18 years

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with essential hypertension being treated in hospitals
Sampling Method: Non-Probability Sample
Enrollment: 2318 (Actual)
Dates: Start 2000-05; Primary Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Change in clinic blood pressure | up to 14 days
Number of patients with adverse drug reactions | up to 14 days